CLINICAL TRIAL: NCT02571218
Title: Substrate-Targeted Catheter Ablation to Treat Persistent Atrial Fibrillation
Brief Title: AF Substrate Mapping and Guided Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SJM-CIP-10054
Record Dates: First submitted 2015-07-27; First posted 2015-10-08 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-04

CONDITIONS: Persistent Atrial Fibrillation
Keywords: atrial fibrillation; mapping; substrate; ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- mCPVA (Active Comparator): Subjects in the mCPVA arm will undergo intervention called "modified circumferential pulmonary vein ablation", which is considered to be the standard ablation treatment for AF.
  Interventions: Device: mCPVA
- Substrate+mCPVA (Experimental): Subjects in the Substrate+mCPVA arm will undergo intervention of substrate mapping and substrate-targeted ablation guided by the investigational device, followed by completion of modified circumferential pulmonary vein ablation.
  Interventions: Device: Substrate+mCPVA

INTERVENTIONS:
Device: Substrate+mCPVA — The intervention in the experimental arm includes using a research software (investigational device) to map AF substrate and guide ablation.
  Arms: Substrate+mCPVA
Device: mCPVA — The intervention in the active comparator arm includes using the commercially available EnSite Velocity mapping and ablation system for modified circumferential pulmonary vein ablation.
  Arms: mCPVA

SUMMARY:
In this study, the investigators aim to identify and characterize, by means of an EnSite Velocity Research Software, the electrophysiological characteristics of substrates that sustain AF in patients with persistent AF and to test whether ablation of such patient-specific substrates might improve the acute and long-term success of conventional catheter ablation therapy.

DETAILED DESCRIPTION:
This study is a prospective, single center, randomized, single-blind, controlled, 2-arm parallel group trial in Milan, Italy.

The total duration of the study is expected to be 24 months with ~12 months of enrollment.

Approximately 80 subjects suffering from persistent AF will be randomized in a 1:1 fashion to the following investigation arms:

* Modified circumferential pulmonary vein ablation alone (mCPVA);
* Substrate-targeted ablation guided by AF substrate mapping, followed by completion of modified circumferential pulmonary vein ablation (Substrate+ mCPVA)

  * Ablate the areas that have fast and regular electrical activities, starting from the fastest cycle length (defined by Mean CL in the range of 120-250 milliseconds, and SD CL in the range of 1-30 milliseconds
  * Ablate the areas that have consistent rotational or focal propagation pattern (defined by conduction velocity vectors)
  * Ablate the areas that comprises the slow conduction zone of possible arrhythmia circuits
  * If AF terminates during RF ablation, stimulation protocol will be used to examine if AF is re-inducible. If AF sustains or is re-inducible and physician decides to remap, mapping will be performed again for substrate-targeted ablation. If AF is not re-inducible, mCPVA will be completed

Subjects will be followed up at 3, 6, 12 months.

The primary objective of the study is to assess acute and long-term outcome of patient-tailored substrate-targeted ablation (Substrate) plus modified circumferential pulmonary vein ablation (Substrate+mCPVA) versus modified circumferential pulmonary vein ablation alone (mCPVA). The secondary objective of the study is to map and characterize electrophysiological substrates during AF, including regular and fast activities, complex fractionated electrograms, wave front propagation directions, and fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 85 years of age
* Persistent AF scheduled to undergo catheter ablation with approved standard indication by ESC/EHRA guidelines
* First or second time ablation for persistent AF
* Ability to provide written informed consent for study participation and be willing and able to comply with the study evaluations and follow up schedule

Exclusion Criteria:

* Had two or more previous AF ablation procedures
* Secondary AF
* Hyperthyroidism
* Left ventricular ejection fraction <30%
* NYHA functional class IV
* Left atrial area > 35 cm2
* Uncorrected severe valvular heart disease
* Contraindication to anticoagulation
* Presence of left atrial thrombus
* Recent (<6 Months) myocardial Infarction or unstable angina or coronary artery by-pass
* Thoracic surgery for congenital, valvular or aortic disease
* History of cerebrovascular accidents
* Pregnancy
* Significant comorbidities such as cancer, severe renal insufficiency requiring hemodialysis, severe obstructive lung disease, cirrhosis, with a life expectancy less than 2 years

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-07; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Pappone, MD, PhD, Principal Investigator — I.R.C.C.S. Policlinico San Donato
Locations (1):
- I.R.C.C.S. Policlinico San Donato, San Donato Milanese, MI, Italy

REFERENCES:
- [Derived] Pappone C, Ciconte G, Vicedomini G, Mangual JO, Li W, Conti M, Giannelli L, Lipartiti F, McSpadden L, Ryu K, Guazzi M, Menicanti L, Santinelli V. Clinical Outcome of Electrophysiologically Guided Ablation for Nonparoxysmal Atrial Fibrillation Using a Novel Real-Time 3-Dimensional Mapping Technique: Results From a Prospective Randomized Trial. Circ Arrhythm Electrophysiol. 2018 Mar;11(3):e005904. doi: 10.1161/CIRCEP.117.005904. PMID 29535136

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | mCPVA | Substrate+mCPVA
Started | 40 | 41
Completed | 40 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | mCPVA | Substrate+mCPVA | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (10.8) | 63.5 (10.4) | 61.7 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 31 | 29 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 40 | 41 | 81
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 40 | 41 | 81
Hypertenstion, n [Count of Participants; unit: Participants] | 26 | 22 | 48
Diabetes mellitus, n [Count of Participants; unit: Participants] | 4 | 4 | 8
Years AF diagnosed, y [Least Squares Mean (Standard Deviation); unit: years] | 3.8 (5.4) | 5.4 (5.3) | 4.5 (5.3)
AF persistency, mo [Mean (Standard Deviation); unit: months] | 6.5 (1.8) | 5.8 (1.3) | 6.1 (1.4)
Left Ventricle Ejection Fraction (%) [Mean (Standard Deviation); unit: %] | 53.5 (5.7) | 55.5 (7.3) | 54.6 (6.6)
LA area, cm2 [Mean (Standard Deviation); unit: cm2] | 24.8 (4.8) | 24.5 (6.1) | 24.5 (5.5)

OUTCOME MEASURES:

1. Primary Outcome: Long-term Clinical Success Rate
Description: Freedom from symptomatic AF off antiarrhythmic drug therapy assessed from the end of the 3 months blanking period to 12 months following the ablation procedure, documented by implantable loop recorder (ILR) monitoring or trans-telephonic (TT) ECG monitoring.
Time Frame: 12 months
Population: Success rate of patient's undergoing radiofrequency catheter ablation during follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | mCPVA | Substrate+mCPVA
Number analyzed (Participants) | 40 | 41
Participants | 30 | 21

2. Secondary Outcome: Acute Ablation Procedure Outcome
Description: Acute AF termination or significant AF cycle length slowing during RF application in ablation procedure
Time Frame: During Ablation
Population: Success rate of radiofrequency catheter ablation to terminate atrial fibrillation during the ablation procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | mCPVA | Substrate+mCPVA
Number analyzed (Participants) | 40 | 41
Participants | 12 | 25

ADVERSE EVENTS:
Time Frame: 1 year throughout the follow up of the study.
Description: Adverse event and or serious adverse event definition does not differ from the clinicaltrials.gov definition.
Arm/Group | mCPVA | Substrate+mCPVA
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/41
Other Adverse Events (participants affected / at risk) | 0/40 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-11): https://cdn.clinicaltrials.gov/large-docs/18/NCT02571218/Prot_SAP_000.pdf